CLINICAL TRIAL: NCT00003997
Title: Phase I Study of MGI-114 (NSC#683863) in Patients With Refractory Myelodysplastic Syndromes, Acute Leukemia and Chronic Myelogenous Leukemia in Blastic Phase (CML-BP)
Brief Title: 6-Hydroxymethylacylfulvene in Treating Patients With Refractory Myelodysplastic Syndrome, Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, or Blastic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02309; MDA-ID-99060; NCI-T99-0043; CDR0000067207 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2001-01

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; blastic phase chronic myelogenous leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — irofulven

ARMS (1):
- Arm I (Experimental): Patients receive 6-hydroxymethylacylfulvene (HMAF) IV over 5 minutes on days 1-5. Treatment repeats every 3-4 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3 patients receive escalating doses of HMAF. The maximum tolerated dose is defined as the dose at which dose limiting toxicity occurs in at least 40% of patients.
  Interventions: Drug: irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
Phase I trial to study the effectiveness of 6-hydroxymethylacylfulvene in treating patients who have refractory myelodysplastic syndrome, acute myeloid leukemia, acute lymphocytic leukemia, or blastic phase chronic myelogenous leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the maximum tolerated dose for 6-hydroxymethylacylfulvene in patients with refractory myelodysplastic syndrome, acute myeloid leukemia, acute lymphocytic leukemia, or blastic phase chronic myelogenous leukemia.

II. Determine the qualitative and quantitative toxicities of this treatment in these patients.

III. Determine the duration and reversibility of the qualitative and quantitative toxicities of this treatment in these patients.

IV. Evaluate, in a preliminary manner, the antileukemic activity of this treatment in these patients.

V. Assess relative mRNA levels of selected NER genes (ERCC1, ERCC2, and ERCC3) in tumor tissues of patients treated with this regimen and correlate with clinical outcome.

OUTLINE: This is a dose escalation study.

Patients receive 6-hydroxymethylacylfulvene (HMAF) IV over 5 minutes on days 1-5. Treatment repeats every 3-4 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3 patients receive escalating doses of HMAF. The maximum tolerated dose is defined as the dose at which dose limiting toxicity occurs in at least 40% of patients.

Patients are followed every 3 months for 1 year and then every 6 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of refractory myelodysplastic syndrome (MDS), acute myeloid leukemia (AML), acute lymphocytic leukemia, or blastic phase chronic myelogenous leukemia MDS and AML include:

  * First salvage with primary refractory disease or first complete remission of no more than 12 months
  * Second or greater salvage
* After the maximum tolerated dose is determined, AML patients with an intermediate prognosis (i.e., complete remission of more than 12 months, but less than 24 months) are eligible
* No candidates for curative therapies such as allogeneic bone marrow transplantation

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: Zubrod 0-2
* Bilirubin no greater than 1.5 mg/dL
* Creatinine no greater than 1.5 mg/dL OR creatinine clearance at least 60 mL/min
* No active congestive heart failure
* No uncontrolled angina
* No myocardial infarction within past 6 months
* No concurrent grade 4 infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No overt psychosis, mental disability, or other incompetency that would preclude obtaining informed consent
* No life threatening nonmalignant illness

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior biologic therapy and recovered
* No concurrent systemic anticancer biologic therapy
* At least 2 weeks since other prior chemotherapy and recovered
* Concurrent hydroxyurea allowed if needed to control blast counts
* No concurrent systemic anticancer chemotherapy
* At least 2 weeks since prior endocrine therapy and recovered
* Concurrent corticosteroids allowed if needed to control blast counts
* At least 2 weeks since prior radiotherapy and recovered
* No concurrent systemic radiotherapy
* No concurrent surgery
* At least 3 weeks since other prior investigational drugs (including analgesics or antiemetics) and recovered
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1999-07; Primary Completion 2000-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis J. Giles, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States